CLINICAL TRIAL: NCT05129007
Title: Pain Monitoring of Herniated Disc Surgery Patients With Oura Ring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Oura health oy (Unknown)
Responsible Party: Sponsor
Other Study IDs: R21071L
Record Dates: First submitted 2021-09-17; First posted 2021-11-22 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Pain Measurement
Keywords: Pain; Oura ring; Activity measurment; Herniated disc
MeSH Terms: conditions — Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All patients
  Interventions: Device: Oura ring

INTERVENTIONS:
Device: Oura ring — Photopletysmography based noninvasive device
  Other Names: Pain questionnaire, BDI-questionnaire

SUMMARY:
The objective of this research study is to show whether data given by Oura ring could be used to objectively measure patients pain and well-being before and after disc surgery.

DETAILED DESCRIPTION:
The study will consist of a total 30 disc prolapse patients. Patients are given Oura rings along with other treatment. Patients use Oura rings before and after disc surgery. Patients will also fill Beck Depression Inventory (BDI) and pain detect inquiries in the beginning and in the end of study. Patients symptoms will also be followed daily by electrical symptom diary.

Oura rings technology is based on photoplethysmography( PPG). PPG is a noninvasive method to detect blood volume changes in the microvascular bed of tissue. PPG waveform varies by respiration, sympathetic nervous system activity and thermoregulation. Oura ring gives information of patients activity level, calorie consumption, steps count, resting heart rate,heart rate variability, respiration rate, body temperature, sleep depth and quality of sleep.

Data collected with Oura ring after disc surgery will be compared to data collected before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Upcoming herniated disc surgery, ability to give a written informed concent

Exclusion Criteria:

* Sleep apnea, Condition with irregular heart rate, lack of cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients from Finland
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate variability | comparison of mean value prior to surgery and one month after surgery
  collected from Oura ring
Change in resting mean heart rate | comparison of mean value prior to surgery and one month after surgery
  collected from Oura ring
Change in ventilatory rate | comparison of mean value prior to surgery and one month after surgery
  collected from oura ring
Change in sleep onset latency | comparison of mean value prior to surgery and one month after surgery
  collected from oura ring
Change in sleep efficiency | comparison of mean value prior to surgery and one month after surgery
  percentage of the time spent asleep while in bed collected from oura ring
Change in number of nighttime awakenings | comparison of mean value prior to surgery and one month after surgery
  collected from oura ring
Change in total sleep time | comparison of mean value prior to surgery and one month after surgery
  collected from oura ring
Change in sleep stages (awake, light sleep, deep sleep and rem sleep) | comparison of mean value prior to surgery and one month after surgery
  percentages of each sleep stages collected from oura ring
Change in symptoms based on symptom diary | prior surgery and one month after surgery
  Daily symptom diary kept by patient

SECONDARY OUTCOMES:
Change in BDI questionnaire points | one month prior surgery and one month after surgery
  BECK Depression Inventory (Scale 1-63, higher scores mean a worse outcome)
Change in pain questionnaire | one month prior surgery and one month after surgery
  Descriptive questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere university hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No